CLINICAL TRIAL: NCT01438099
Title: Reliability of Ultrasound Assisted Epidural Analgesia in Obese and Normal Weight Parturients
Status: Completed | Type: Observational
Sponsor: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Paolo Severgnini, Prof., Università degli Studi dell'Insubria
Other Study IDs: 18894
Record Dates: First submitted 2011-09-14; First posted 2011-09-21 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2013-08

CONDITIONS: Pregnancy
Keywords: epidural analgesia; ultrasound; labor analgesia; labor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- normal subjects: parturients admitted to the labor ward who request epidural analgesia with BMI < 30
- obese subjects: parturients admitted to the labor ward who request epidural analgesia with BMI > 30

SUMMARY:
This study wants to investigate if ultrasound assisted epidural catheter insertion for labor analgesia is easier and safer to the standard epidural technique.

DETAILED DESCRIPTION:
This study has four specific aims:

1. to evaluate congruity between palpatory technique and ultrasound lumbar evaluation to identify the correct spinal space;
2. to compare between ultrasound evaluation and needle measure of skin-epidural space depth;
3. to compare between longitudinal and transverse ultrasound epidural space depth in obese and normal parturients;
4. to check the reduction of complications and failure rates of epidural analgesia with ultrasound assistance.

ELIGIBILITY:
Inclusion Criteria:

* all women who request epidural analgesia for labor

Exclusion Criteria:

* all women who present contraindication for epidural analgesia

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: all women after thirty weeks of pregnancy, experiencing spontaneous or induced labor
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2011-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
The congruity between palpatory technique and ultrasound lumbar evaluation | participants will be followed for the duration of hospital stay, an expected average of 3 days
  The congruity between palpatory technique and ultrasound lumbar evaluation to identify the correct spinal space performing epidural analgesia

SECONDARY OUTCOMES:
Longitudinal and transverse ultrasound epidural space depth in obese and normal parturients | participants will be followed for the duration of hospital stay, an expected average of 3 days
  Longitudinal and transverse ultrasound epidural space depth in obese and normal parturients will be measured and compared to the needle depth

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Severgnini, Prof., Principal Investigator — Universita' degli Studi dell'Insubria, Varese, Italy
Locations (1):
- Azienda ospedaliera ospedale Circolo e Fondazione Macchi, Varese, Varese, Italy